CLINICAL TRIAL: NCT06734767
Title: The Effect of an MBSR Course on Medical Trainee and Medical Academic Faculty Stress and Burnout
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jeffrey Zahn, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STUDY-23-01113
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Burnout
Keywords: Burnout; MBSR; mindfulness; physician well-being
MeSH Terms: conditions — Burnout, Psychological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Medical practitioners who choose to register for a free mindfulness course are evaluated for improvements in their ability to manage stress and mitigate burnout.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Course participants are offered to enroll anonymously in this survey study and are unaware of the who the study results reviewers will be.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness Based Stress Reduction course faculty participants (Other): Faculty physicians who have chosen to take the free 8-week course are offered the opportunity to anonymously enroll in the study.
  Interventions: Behavioral: Mindfulness Based Stress Reduction 8-week course
- Mindfulness Based Stress Reduction course trainee participants (Other): Trainee physicians who have chosen to take the free 8-week course are offered the opportunity to anonymously enroll in the study.
  Interventions: Behavioral: Mindfulness Based Stress Reduction 8-week course

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction 8-week course — The Mindfulness Based Stress Reduction (MBSR) 8-week course is an evidence-based curriculum that has been taught for over 40 years and is offered world-wide, teaching mindfulness skills and practices such as meditation.

SUMMARY:
The study team is seeking to evaluate the efficacy of the Mindfulness Based Stress Reduction (MBSR) course at reducing stress and burnout. This will be done through the collection of brief anonymous online surveys (the Perceived Stress Scale and the Mini Z) before the MBSR course and at 2 weeks, 6 months, and 12 months following the end of the course. Participation is completely voluntary and will not affect anyone's ability to take this course, and the course instructors will have no knowledge of who has or has not participated in the study.

DETAILED DESCRIPTION:
The study is a pre- and post- survey design with the 8-week MBSR course as the intervention. MBSR is an evidence-based curriculum with a greater than 40-year history, that has been taught at Mount Sinai since 2018. Study participants will be those who have voluntarily signed up to take the course in response to an email describing the course that was sent by the office of the Mount Sinai Graduate Medical Education (GME). The study participants will be separated into two groups: faculty and trainees, and the study will span approximately two weeks prior to the start of the course (9/13/2023) (the "pre-" period) and six months after the completion of the course 5/31/2024) (the "post-" period). The course will be delivered by Zoom, but the participants will be joining from all Mount Sinai locations. The MBSR course itself involves didactics (i.e., stress physiology, review of mindfulness research, mindful communication practices), group discussions based on individual experiences with the mindful practices taught in the course, and the teaching of meditation practices including sitting and moving meditation practices. Home practices are offered as guidance each week but are not required. There is no planned control group at this time.

ELIGIBILITY:
Inclusion Criteria:

- A physician in The Mount Sinai Hospital System

Exclusion Criteria:

- none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | Baseline and at 2 weeks, 6 months, and 12 months following the end of the course (course is 8 weeks)
  The Perceived Stress Scale (PSS) is a validated 10-question survey tool that evaluates an individual's stress level. Each question is scored from 0-4 - Full scale range from 0-40, with higher score indicating higher perceived stress.

SECONDARY OUTCOMES:
The "Mini Z" survey | Baseline and at 2 weeks, 6 months, and 12 months following the end of the course (course is 8 weeks)
  The Mini Z is a validated one-question survey designed to gauge the degree of burnout an individual is experiencing.
  Full score from 1-5, with higher score indicating more burnout.
Burnout questions | Baseline and at 2 weeks, 6 months, and 12 months following the end of the course (course is 8 weeks)
  How often do you feel "burned out' by your work? How often do you feel you've become more callous toward people since you took this job? Each question is scored 0-6, with cumulate total score from 0-12. Higher score indicates more burnout.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Zahn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Surveys are filed anonymously, no identifying information of participants